CLINICAL TRIAL: NCT00465452
Title: The Impact of Switching to Continuous Release Dopamine Agonists on Non-Motor Side Effects
Brief Title: Impact of Switching to Continuous Release Dopamine Agonists
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Toledo (Other)
Responsible Party: Principal Investigator, Lawrence Elmer, MD, PhD, Professor, Med Dir, Cntr for Neurological Disorders, University of Toledo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MUO-04
Record Dates: First submitted 2007-04-24; First posted 2007-04-25 (Estimated); Results first posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Continuous Release Dopamine Agonists (Experimental): Continuous Release Dopamine Agonists
  Interventions: Drug: Continuous Release Dopamine Agonists

INTERVENTIONS:
Drug: Continuous Release Dopamine Agonists — Continuous Release Dopamine Agonists
  Other Names: ropinirole extended release

SUMMARY:
The purpose of this proposal is to determine if switching PD patients treated with pramipexole to ropinirole CR reduces the non-motor side effects frequently experienced by these patients. Side effects that we will monitor in particular include somnolence, peripheral edema, cognitive decline with and without hallucinations. PD patients followed in the MUO Neurology Clinic who are being treated with pramipexole and have evidence of at least one of the following symptoms: somnolence, cognitive impairment with or without hallucinations, or peripheral edema will be offered the opportunity to participate in this study.

DETAILED DESCRIPTION:
The purpose of this proposal is to determine if switching PD patients treated with pramipexole to ropinirole CR reduces the non-motor side effects frequently experienced by these patients. Side effects that we will monitor in particular include somnolence, peripheral edema, cognitive decline with and without hallucinations. PD patients followed in the MUO Neurology Clinic who are being treated with pramipexole and have evidence of at least one of the following symptoms: somnolence, cognitive impairment with or without hallucinations, or peripheral edema will be offered the opportunity to participate in this study.

Fifteen subjects who are currently receiving pramipexole therapy (monotherapy or adjunctive therapy) who are experiencing one or more of the following symptoms: somnolence, cognitive decline with/without hallucinations, and peripheral edema will be asked if they are willing to participate at the time of their clinic visit at the PDMDP.

The crossover from pramipexole to ropinirole CR will be performed over a 2 week interval. During the first week, the initial drug dose will substitute ½ of the pramipexole with ½ of the target dose of ropinirole CR. If subjects are tolerating the drug change, then 100% of the target dose of ropinirole CR (and no pramipexole) will be started in the second week.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet all of the following inclusion criteria to qualify for entrance into the study:

* Subjects who are male or female and are aged 55 and older.
* Subjects and/or their legal guardians must be able and willing to give informed consent.
* Subjects must be on stable doses of pramipexole for greater than 4 weeks duration prior to screening.
* Subjects who are female must be non-pregnant and non-nursing. Women of Child-Bearing Potential (WOCBP) must use a reliable method of contraception (e.g., oral contraceptive or long-term injectable or implantable hormonal contraceptive, double-barrier methods, such as condom and diaphragm, condom and foam, condom and sponge or intra-uterine devices) and have a negative serum pregnancy test at screening. Women are considered to not be of child-bearing potential if they have been surgically sterilized (physician-documented hysterectomy or tubal ligation) or if they are post-menopausal.
* Subjects must have a clinical diagnosis of Parkinson's based on the presence of at least 2 of the 3 cardinal criteria - rest tremor, bradykinesia, rigidity - and no obvious history of head trauma, stroke, infectious, structural, or metabolic abnormality consistent with an alternative diagnosis to Parkinson's disease.
* Evidence of one or more of the following symptoms: somnolence (ESS score ≥ 9), cognitive decline (MMSE < 24 ± presence of hallucinations (NPI-Q), peripheral edema (present by objective physical exam with baseline ankle and calf circumference measured in centimeters).

Exclusion Criteria:

A subject who meets any of the following criteria will NOT qualify for the study:

* Subjects must not be receiving any treatments for excess somnolence such as amphetamine derivatives, other stimulants or Provigil.
* Subjects with actively treated malignancies, clinically significant heart disease, kidney, liver, or pulmonary disorders will be excluded.
* Subjects with clinical depression who are not receiving stable doses of antidepressant therapy in excess of 4 weeks duration.
* Subjects with history of orthostatic hypotension (>30mm drop in systolic pressure and/or >20mm drop in diastolic pressure) associated with syncope.
* Subjects started within the last 14 days on any drug known to substantially inhibit CYP1A2 (e.g., cimetidine, fluvoxamine) or induce CYP1A2 (e.g.omeprazole) (Note: Subjects already on these agents may be enrolled but must remain on the stable doses of the agents from 14 days prior to the beginning of the study).
* Subjects who have other medical conditions that are considered clinically unstable or that may compromise the safety of the patient during this study.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-01; Primary Completion 2009-03 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Elmer, MD, PhD, Principal Investigator — Medical University of Ohio
Locations (1):
- Medical University of Ohio, Toledo, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients from our outpatient clinic with Parkinson's disease receiving regular pramipexole as one of their treatments and experiencing one or more of the side effects measured in this study.
Groups:
- Continuous Release Dopamine Agonists: Patients were switched from regular pramipexole to extended release ropinirole
Period: Overall Study
Arm/Group | Continuous Release Dopamine Agonists
Started | 11
Completed | 10
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Continuous Release Dopamine Agonist: Patients were switched from regular pramipexole to extended release ropinirole
Arm/Group | Continuous Release Dopamine Agonist
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] — years at entry into study
  years | 58 (8.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS), Parts 3 (Motor Performance) and 4 (Disability).
Description: The Unified Parkinson's Disease Rating Scale (UPDRS), parts 3 (motor performance) and 4 (disability) are standardized and validated measures of various symptoms of Parkinson's disease - total scores range from 0 to 148 with lower scores representing better Parkinson symptom control and higher scores representing worse symptoms of Parkinson's.
Time Frame: initial visit and at end of study 24 weeks
Population: Patients with Parkinson's disease receiving regular pramipexole as one of their treatments and experiencing one or more of the side effects measured in this study.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Continuous Release Dopamine Agonist
Number analyzed (Participants) | 10
score on a scale
  UPDRS Part 3 Baseline | 19.2 [0 to 108]
  UPDRS Part 3 Week 24 | 17.6 [0 to 108]
  UPDRS Part 4 Baseline | 5.1 [0 to 24]
  UPDRS Part 4 Week 24 | 2.9 [0 to 24]

2. Primary Outcome: Mini-Mental Status Exam (MMSE), the Clock Drawing Test (CDT), the Patient Health Questionnaire (PHQ-9).
Description: The Mini-Mental Status Exam (MMSE) and the Clock Drawing Test (CDT) are standardized and validated measures of cognitive function. The Patient Health Questionnaire (PHQ-9) is a standardized and validated measure of quality of life. The Mini-Mental Status Exam (MMSE) scale is 0-30 with higher numbers indicating improvement. The Clock Drawing Test (CDT) range is 0-10 with higher numbers indicating improvement. the PHQ scale is 0-27 with lower numbers indicating improved outcome.
Time Frame: initial visit and at end of study 24 weeks
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Continuous Release Dopamine Agonists: This group was switched from regular pramipexole to extended release ropinirole.
Arm/Group | Continuous Release Dopamine Agonists
Number analyzed (Participants) | 10
score on a scale
  MMSE Baseline | 28.9 [0 to 30]
  MMSE 24 Weeks | 29.1 [0 to 30]
  Clock Drawing Test Baseline | 9.8 [0 to 10]
  Clock Drawing Test 24 Weeks | 9.4 [0 to 10]
  Patient Health Questionnaire Baseline | 7.5 [0 to 27]
  Patient Health Questionnaire Week 24 | 6.2 [0 to 27]

3. Primary Outcome: Peripheral Edema, as Measured by Quantitative Assessment of Ankle Edema
Description: The assessment of ankle edema was considered to be a marker of improvement possibly seen in patients who switched from regular pramipexole to extended release ropinirole. .
Time Frame: initial visit and at end of study 24 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: mm
Groups:
- Continuous Release Dopamine Agonist: Subjects were switched from regular pramipexole to extended release ropinirole
Arm/Group | Continuous Release Dopamine Agonist
Number analyzed (Participants) | 10
mm
  Ankle Edema Baseline | 225.11 [207.7 to 265.2]
  Ankle Edema Week 24 | 224.38 [203.6 to 262.7]

4. Primary Outcome: Patient Satisfaction Questionnaire
Description: The patient satisfaction/preference (Patient Satisfaction Questionnaire - PS) scores vary from 0-10 with higher scores indicating greater satisfaction with the med change.
Time Frame: initial visit and at end of study 24 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Continuous Release Dopamine Agonist
Number analyzed (Participants) | 10
score on a scale
  Patient Satisfaction Questionnaire Baseline | 0.7 [0 to 10]
  Patient Satisfaction Questionnaire Week 24 | 5.2 [0 to 10]

5. Primary Outcome: Parkinson's Disease Questionnaire (PDQ-39)
Description: The Improvement in quality of life (Parkinson's Disease Questionnaire - PDQ-39 - is a standardized and validated measure of patient quality of life ranging in score from 0-100 with lower scores indicating improvement versus higher scores indicating worsening of QOL.
Time Frame: initial visit and at end of study 24 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Continuous Release Dopamine Agonist
Number analyzed (Participants) | 10
score on a scale
  PDQ-39 Baseline | 32.3 [0 to 100]
  PDQ-39 Week 24 | 31.1 [0 to 100]

6. Other Pre Specified Outcome: Epworth Sleepiness Scale (ESS).
Description: Epworth sleepiness scale is a standardized and validated measure of patient's daytime sleepiness. The range of scores is from 0-24 with lower scores representing minimal to no sleepiness and higher scores indicating excessive daytime somnolence.
Time Frame: initial visit and at end of study 24 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Continuous Release Dopamine Agonist: Patients were switched from regular release pramipexole to extended release ropinirole
Arm/Group | Continuous Release Dopamine Agonist
Number analyzed (Participants) | 10
score on a scale
  Epworth sleepiness scale Baseline | 18.2 [0 to 24]
  Epworth sleepiness scale Week 24 | 11.9 [0 to 24]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Continuous Release Dopamine Agonist
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 11/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous Release Dopamine Agonist (N=11)
General pains (General disorders) | 11 (68)
Hypertension (Cardiac disorders) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 7 (10)
Injury (Injury, poisoning and procedural complications) | 3 (6)
Nervous System (Nervous system disorders) | 10 (23)
Increased Compulsion (Psychiatric disorders) | 1 (2)
Upper Respiratory (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Skin (Skin and subcutaneous tissue disorders) | 1 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes